CLINICAL TRIAL: NCT02243189
Title: A Phase 1 Study to Examine the Cytokine Levels, Gene Expression and Safety of a Single Nasal Dose of JNJ-43260295, in a Double-Blind, Randomized, Placebo-Controlled Setting in Healthy Subjects, and by an Open-Label Assessment in Atopic Subjects With Mild to Mild-Persistent Asthma With and Without Nasal Allergen Challenge Prior to Dosing
Brief Title: Study to Examine the Cytokine Levels, Gene Expression and Safety of a Single Nasal Dose of JNJ-43260295, in Healthy Participants, and Atopic Participants With Mild to Mild-Persistent Asthma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Under enrollment and IP supply expiring.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR105491; 43260295HRV1003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-09-16; First posted 2014-09-17 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Healthy; Asthma
Keywords: Healthy; Asthma; JNJ-43260295; Nasal Allergen Challenge
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- JNJ-43260295 (Healthy Participants) (Experimental): Participants will receive a single nasal dose of JNJ-43260295, 6400 microgram, equally spread over the two nostrils.
  Interventions: Drug: JNJ-43260295
- Placebo (Healthy Participants) (Placebo Comparator): Participants will receive a single nasal dose of placebo matching to JNJ-43260295.
  Interventions: Drug: Placebo
- JNJ-43260295 (Asthmatic Participants) (Experimental): Participants will participate in 3 consecutive treatment periods (Periods 1, 2, and 3). In Period 1, each participant will receive a single nasal dose of JNJ-43260295 without prior nasal allergen challenge. In Period 2, each participant will receive a single nasal dose of JNJ-43260295, preceded by a nasal allergen challenge approximately 15 hours prior to the dosing. In Period 3, each participant will receive single nasal allergen challenge without JNJ-43260295. There will be a washout period of at least 21 days between 3 consecutive treatment periods.
  Interventions: Drug: JNJ-43260295; Drug: Nasal Allergen Challenge

INTERVENTIONS:
Drug: JNJ-43260295 — A single nasal dose of JNJ-43260295, 6400 microgram, will be given.
  Arms: JNJ-43260295 (Asthmatic Participants); JNJ-43260295 (Healthy Participants)
Drug: Placebo — A single nasal dose of placebo matching to JNJ-43260295 will be given.
  Arms: Placebo (Healthy Participants)
Drug: Nasal Allergen Challenge — Participants will be challenged by the nasal route with an appropriate allergen based on skin test reactivity.
  Arms: JNJ-43260295 (Asthmatic Participants)

SUMMARY:
The purpose of this study is to investigate the cytokine levels in nasal lavage and gene expression in nasal scraping following a single nasal dose of JNJ-43260295 in healthy participants, and in atopic mild to mild-persistent asthmatic (breathing disorder in which there is wheezing and difficulty in breathing) participants with and without nasal allergen challenge prior to dosing.

DETAILED DESCRIPTION:
This study consists of 2 parts. In first part, healthy adult participants will receive a single nasal dose of JNJ-43260295 or placebo in a double blind (both the participant and investigator do not know whether participant is assigned to receive study medication or placebo), randomized (study medication or placebo assigned to participants by chance), and placebo-controlled (study in which the experimental treatment or procedure is compared to a placebo) setting. In second part, which will be open label (participants and investigators are aware about the treatment, participants are receiving), atopic participants with mild to mild-persistent asthma will participate in 3 consecutive treatment periods (Period 1, 2, and 3). In Period 1, each participant will receive a single nasal dose of JNJ-43260295 without prior nasal allergen challenge. In Period 2, each participant will receive a single nasal dose of JNJ-43260295, preceded by a nasal allergen challenge approximately 15 hours prior to the JNJ-43260295 dosing. In Period 3, each participant will receive single nasal allergen challenge without JNJ-43260295. There will be a washout period of at least 21 days between 3 consecutive treatment periods. Cytokine levels in nasal lavage and gene expression in nasal scraping will be primarily evaluated during all treatment periods. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

A. Healthy Participants and Atopic Mild to Mild-Persistent Asthmatic Participants:

* Participants must be non-smokers or non-regular smokers (1 to 2 cigarettes on the weekend as part of social gathering) for at least 3 months prior to Screening, according to the participant's self-reported medical history. Participants should be willing to (continue to) abstain from smoking from Screening until completion of the last study related activity
* Participants must have a body mass index (BMI: weight in kilogram [kg] divided by the height in square meter [m^2]) of 18.0 to 30.0 kg/m^2, extremes included
* Participants must have a normal 12-lead electrocardiogram (ECG) at Screening including normal sinus rhythm (heart rate between 40 and 100 beats per minute [bpm]); QT interval corrected for heart rate according to Fridericia (QTcF) interval less than and equal to (<=) 450 milliseconds (ms); QRS interval lower than 120 ms; and PR interval <=220 ms
* Participants must be healthy, with the exception of findings related to asthma and allergy in atopic mild to mild-Persistent asthmatic participants, on the basis of a medical evaluation that reveals the absence of any clinically relevant abnormality and includes a physical examination, medical history, vital signs (Systolic Blood Pressure [BP], Diastolic BP, pulse rate, respiratory rate, and body temperature), and the results of blood biochemistry and hematology tests performed at Screening
* Participants must be willing/ able to adhere to the prohibitions and restrictions specified in the protocol and study procedures

B. Atopic Mild to Mild-Persistent Asthmatic Participants:

* Participants with Investigator-diagnosed mild to mild-persistent asthma based on the Guidelines for the Diagnosis and Management of Asthma
* Participants having a well-established allergen profile (participants have been previously skin tested and, by history, have allergic responses to specific allergens)
* Participants with forced expiratory volume in 1 second (FEV1) greater than (>) 70 percent (%) of predicted at Baseline

Exclusion Criteria:

A. Healthy Participants and Atopic Mild to Mild-Persistent Asthmatic Participants:

* Participants having a significant (by the assessment of the Investigator) nasal abnormality and/or has a history of nasal or sinus surgery within 12 months of enrollment
* Participants having an upper or lower respiratory tract infection within 4 weeks of enrollment
* Participants with a history or evidence of use of alcohol, barbiturates, amphetamines, recreational or narcotic drug use within the past 1 year, which in the Investigator's opinion would compromise participant's safety and/or compliance with the study procedures
* Participants with a known history of human immunodeficiency virus type 1 (HIV-1) or HIV-2 infection, or with a known history of hepatitis A, B, or C virus infection at study Screening
* Female participants who are breastfeeding at Screening or having a positive urine pregnancy test at Screening

B. Atopic Mild to Mild-Persistent Asthmatic Participants:

* Hospitalization or treatment in an emergency care facility for asthma during the last 3 years
* Participants using nasal corticosteroids on a daily basis in the 4 weeks prior to enrollment
* Participants who have received allergen immunotherapy in the last 2 years

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Cytokine Levels in Nasal Lavage | Up to 48 hours post dose
  Sixteen cytokines will be assessed: interferon alpha (IFN-alpha), IFN-beta, IFN-gamma, IFN-lambda, interleukin-1 alpha (IL-1 alpha), IL-4, IL-5, IL-6, IL 8, IL-10, IL-12p70, IL-13, IL-15, IL-17, IL-23, and tumor necrosis factor-alpha (TNF-alpha), using the 16-plex kit.
Gene Expression in Nasal Scrapings | Up to 48 hours post dose
  Gene expression will be determined by analyzing total ribonucleic acid (RNA) by microarray chips.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs) | AEs: Baseline up to 8 days after the last dose of study drug; SAEs: Baseline up to 30 days after the last dose of study drug
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; or congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Charlottesville, Virginia, United States